CLINICAL TRIAL: NCT03017079
Title: A More Physiological Feeding Process in ICU:the Intermittent Infusion With Semi-solidification of Nutrients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Man Huang, Ph.D, Clinical Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: lukongmiao123
Record Dates: First submitted 2017-01-06; First posted 2017-01-11 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Nutrition, Enteral
Keywords: Semi-solidification; caloric debt; enteral nutrition; critical illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semi-solidification with nutrient (Experimental): semi-solidification with nutrient:after infusion of semi-solid agent, enteral nutrition is applied less than 60 mins.
  Intervention: Other: bolus Intermittent enteral feeding
  Interventions: Dietary Supplement: semi-solid agent with standard enteral feeding
- Standard enteral nutrition (Placebo Comparator): After infusion of Sterile Water for Injection,bolus Intermittent enteral feeding via the nasogastric tube is applied less than 60 mins.
  Intervention: Other: Standard enteral feeding
  Interventions: Other: standard enteral feeding

INTERVENTIONS:
Dietary Supplement: semi-solid agent with standard enteral feeding — after infusion of semi-solid agent, Intermittent enteral feeding is applied less than 60 minutes
  Other Names: semi-solidification of nutrient
  Arms: semi-solidification with nutrient
Other: standard enteral feeding — Intermittent enteral feeding is applied less than 60 minutes
  Other Names: standard enteral nutrition
  Arms: Standard enteral nutrition

SUMMARY:
Malnutrition and underfeeding are major challenges in caring for critically ill patients. Continuous feeding were thought to be better tolerated by patients with the limited absorptive gut surface area or gastrointestinal dysfunction, but associated with more tube clogging and required the patient to be attached to an infusion pump for significant periods of time. Intermittent infusion resembled more physiological feeding process, which allowed greater patient mobility and might reach goal enteral calories earlier, and the latter were considered to effectively decrease the length of stay (LOS)-in-hospital and mortality. However, it also had some previous study found that intermittent infusion had more complications, such as diarrhea, regurgitation than continuous. Some study found that it was an efficient way to prevent aspiration and reflux by increasing the enteral nutrient solution viscosity and improve bolus intermittent feeding intolerance. The primary goal of this was to study whether receiving semi-solidification of nutrients could increase the percent prescribed calories received by improving the feeding intolerance, and secondary goal was to observing the effect of semi-solid nutrient to the LOS of ICU and in-hospital, lung infection, 30-days mortality and the glycemic variability (GV).

DETAILED DESCRIPTION:
Enteral nutrition (EN) therapy is an essential part in critically ill patients，and can be administered on a continuous or intermittent, but there were no consensus on which should be adopted. Continuous feeding were thought to be better tolerated by patients with the limited absorptive gut surface area or gastrointestinal dysfunction, but associated with more tube clogging and required the patient to be attached to an infusion pump for significant periods of time. Intermittent infusion resembled more physiological feeding process, which allowed greater patient mobility and might reach goal enteral calories earlier, and the latter were considered to effectively decrease the LOS-in-hospital and mortality. However, it also had some previous study found that intermittent infusion had more complications, such as diarrhea, regurgitation than continuous.

Recently, some study found that it was an efficient way to prevent aspiration and reflux by increasing the enteral nutrient solution viscosity and improve bolus intermittent feeding intolerance. In dementia or Parkinson's patients, one study showed that high-viscosity liquid meal could decrease the incidence of aspiration, compared with the thin liquid, but the study about the viscosity of nutrition was little and the sample size was small.

In this study, the primary goal of this was to study whether receiving semi-solidification of nutrients could increase the percent prescribed calories received by improving the feeding intolerance, and secondary goal was to observing the effect of semi-solid nutrient to the LOS of ICU and in-hospital, lung infection, 30-days mortality and the glycemic variability (GV).

ELIGIBILITY:
Inclusion Criteria:

(1)14 years and older, who received EN for more than 72 hours, were eligible for inclusion (2) all patients started on EN by nasogastric tube

Exclusion Criteria:

1. received EN <72 hours
2. received EN prior to ICU admission
3. had acute pulmonary infection
4. had history of Gastrointestinal surgery
5. had contraindications of EN, such as intestinal obstruction (mechanical or paralytic ileus).

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: man huang, phD, Principal Investigator — Second affiliated hospital, Zhejiang university school of medicine
Locations (1):
- Second affiliated hospital, Zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peev MP, Yeh DD, Quraishi SA, Osler P, Chang Y, Gillis E, Albano CE, Darak S, Velmahos GC. Causes and consequences of interrupted enteral nutrition: a prospective observational study in critically ill surgical patients. JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):21-7. doi: 10.1177/0148607114526887. Epub 2014 Apr 7. PMID 24714361
- [Result] Evans DC, Forbes R, Jones C, Cotterman R, Njoku C, Thongrong C, Tulman D, Bergese SD, Thomas S, Papadimos TJ, Stawicki SP. Continuous versus bolus tube feeds: Does the modality affect glycemic variability, tube feeding volume, caloric intake, or insulin utilization? Int J Crit Illn Inj Sci. 2016 Jan-Mar;6(1):9-15. doi: 10.4103/2229-5151.177357. PMID 27051616
- [Result] MacLeod JB, Lefton J, Houghton D, Roland C, Doherty J, Cohn SM, Barquist ES. Prospective randomized control trial of intermittent versus continuous gastric feeds for critically ill trauma patients. J Trauma. 2007 Jul;63(1):57-61. doi: 10.1097/01.ta.0000249294.58703.11. PMID 17622869
- [Result] Taylor BE, McClave SA, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society of Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). Crit Care Med. 2016 Feb;44(2):390-438. doi: 10.1097/CCM.0000000000001525. No abstract available. PMID 26771786
- [Result] Logemann JA, Gensler G, Robbins J, Lindblad AS, Brandt D, Hind JA, Kosek S, Dikeman K, Kazandjian M, Gramigna GD, Lundy D, McGarvey-Toler S, Miller Gardner PJ. A randomized study of three interventions for aspiration of thin liquids in patients with dementia or Parkinson's disease. J Speech Lang Hear Res. 2008 Feb;51(1):173-83. doi: 10.1044/1092-4388(2008/013). PMID 18230864
- [Result] Bardhan KD, Strugala V, Dettmar PW. Reflux revisited: advancing the role of pepsin. Int J Otolaryngol. 2012;2012:646901. doi: 10.1155/2012/646901. Epub 2011 Nov 10. PMID 22242022
- [Result] Hayat JO, Gabieta-Somnez S, Yazaki E, Kang JY, Woodcock A, Dettmar P, Mabary J, Knowles CH, Sifrim D. Pepsin in saliva for the diagnosis of gastro-oesophageal reflux disease. Gut. 2015 Mar;64(3):373-80. doi: 10.1136/gutjnl-2014-307049. Epub 2014 May 7. PMID 24812000
- [Derived] Lu K, Zeng F, Li Y, Chen C, Huang M. A more physiological feeding process in ICU: Intermittent infusion with semi-solid nutrients (CONSORT-compliant). Medicine (Baltimore). 2018 Sep;97(36):e12173. doi: 10.1097/MD.0000000000012173. PMID 30200118

RESULTS

PARTICIPANT FLOW:
Groups:
- Semi-solidification With Nutrient: semi-solidification with nutrient:after infusion of semi-solid agent, enteral nutrition is applied less than 60 mins.
  Intervention: Other: bolus Intermittent enteral feeding
  semi-solid agent: after infusion of semi-solid agent, Intermittent enteral feeding is applied less than 60 mins
- Standard Enteral Nutrition: After infusion of Sterile Water for Injection,bolus Intermittent enteral feeding via the nasogastric tube is applied less than 60 mins.
  Intervention: Other: Standard enteral feeding
  standard enteral feeding: Intermittent enteral feeding is applied less than 60 mins
Period: Overall Study
Arm/Group | Semi-solidification With Nutrient | Standard Enteral Nutrition
Started | 20 | 20
Completed (Death:defined as death within 3 days of enrollment) | 14 | 14
Not Completed | 6 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Death | 3 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semi-solidification With Nutrient | Standard Enteral Nutrition | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.93 (20.96) | 52.14 (13.77) | 53.54 (17.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 14 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 14 | 14 | 28
NRS 2002 [Mean (Standard Deviation); unit: units on a scale] — NRS 2002 range from 0 to 7,and The higher the score, the higher the nutritional risk
  units on a scale | 3.14 (0.77) | 2.86 (0.95) | 3 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: the Ratio of the Enteral Nutrition
Description: the ratio of the enteral nutrition=administered volume of enteral nutrition / prescribed volume of nutrition X 100%; This ratio fluctuates between 0 and 100%, and the higher the ratio, the higher the execution rate
Time Frame: 3 days after receiving enteral nutrition
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Intermittent Feeding With Semi-solid Nutrients: semi-solidification with nutrient:after infusion of semi-solid agent, enteral nutrition is applied less than 60 mins.
- Standard Enteral Feeding: After infusion of Sterile Water for Injection,bolus Intermittent enteral feeding via the nasogastric tube is applied less than 60 mins.
  Intervention: Other: Standard enteral feeding
  standard enteral feeding: Intermittent enteral feeding is applied less than 60 mins
Arm/Group | Intermittent Feeding With Semi-solid Nutrients | Standard Enteral Feeding
Number analyzed (Participants) | 14 | 14
ratio | 0.98 (0.067) | 0.73 (0.15)

2. Secondary Outcome: the Patient of Feeding Intolerance（FI）
Description: the definition of FI was included one of the conditions:diarrhea, vomiting, regurgitation, obvious bowel distension and GRV>200mL.
  Due to the small sample size, only the number of patients who occurred was recorded.
Time Frame: 3 days
Measure: Number; unit: participants
Groups:
- Intermittent Feeding: After infusion of Sterile Water for Injection,bolus Intermittent enteral feeding via the nasogastric tube is applied less than 60 mins.
  Intervention: Other: Standard enteral feeding
  standard enteral feeding: Intermittent enteral feeding is applied less than 60 mins
- Intermittent Feeding With Semi-solid Nutrients: semi-solidification with nutrient:after infusion of semi-solid agent, enteral nutrition is applied less than 60 mins.
  Intervention: Other: bolus Intermittent enteral feeding
  semi-solid agent: after infusion of semi-solid agent, Intermittent enteral feeding is applied less than 60 mins
Arm/Group | Intermittent Feeding | Intermittent Feeding With Semi-solid Nutrients
Number analyzed (Participants) | 14 | 14
participants | 8 | 2
Statistical Analysis 1: Comparison: Intermittent Feeding; P=.046; Test type: Non-Inferiority — a:0.05;β：0.01 P=.046; p = 0.05, t-test, 2 sided

3. Secondary Outcome: the Patients With Lung Infection
Description: patient contain the following three conditions:
  1.Sputum volume increased or Sputum properties change;2.CT Scan-Chest suggest that there was lung infection; 3.CRP and / or PCT increased
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Intermittent Feeding | Intermittent Feeding With Semi-solid Nutrients
Number analyzed (Participants) | 14 | 14
participants | 8 | 7
Statistical Analysis 1: Comparison: Intermittent Feeding vs Intermittent Feeding With Semi-solid Nutrients; Test type: Non-Inferiority — a 0.05; p = 0.05, t-test, 2 sided; Odds Ratio (OR) = 0.05

4. Secondary Outcome: 30-days Mortality
Description: dead within 30 days in ICU
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Intermittent Feeding: After infusion of Sterile Water for Injection,bolus Intermittent enteral feeding via the nasogastric tube is applied less than 60 mins.
Arm/Group | Intermittent Feeding With Semi-solid Nutrients | Intermittent Feeding
Number analyzed (Participants) | 14 | 14
participants
  The number of deaths within 30 days after ICU | 3 | 2
  The number of live after 30 days in ICU | 11 | 12
Statistical Analysis 1: Comparison: Intermittent Feeding With Semi-solid Nutrients; Test type: Superiority; p = 0.05, Chi-squared, Corrected

5. Secondary Outcome: the Glycemic Variability(GV)
Description: Divided into three grades:I:GV less than 4mmol/24h; II 4-6mmol/24h;III more than 6mmol/24h
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mmol/l
Groups:
- Intermittent Feeding With Semi-solid Nutrients: the initial feeds of 100 to 300mL every 4 to 8 hours and the semi-solid agent feeded before the EN application within 1 hour, which is low methoxy pectin gel and water-soluble dietary fiber form apple and citrus peel by binding to calcium ions in EN to increase the viscosity, but do not change any chemical properties of EN. This was repeated twice and, if tolerated, they were advanced by 100 to 300mL every 1 to 2 days to the volume goal.
- Intermittent Feeding: The intermittent protocol involved initial feeds of 100 to 300mL every 4 to 8hours. This was repeated twice and, if tolerated, they were advanced by 100 to 300mL every 1 to 2 days to the volume goal. Each intermittent feeding was delivered via an enteral feeding pump during a 30- to 60-minute period of time.
Arm/Group | Intermittent Feeding With Semi-solid Nutrients | Intermittent Feeding
Number analyzed (Participants) | 14 | 14
mmol/l
  1d-0h | 7.514 (2.2309) | 8.457 (2.9456)
  1d-4h | 8.336 (2.1653) | 9.700 (3.1001)
  1d-8h | 9.229 (3.2587) | 9.664 (3.1023)
  1d-12h | 9.342857 (3.1353357) | 8.985714 (3.2846630)
  1d-16h | 8.635714 (2.4069154) | 8.992857 (3.1086639)
  1d-20h | 8.064286 (1.9727400) | 8.721429 (2.5137097)
  2d-0h | 8.436 (2.2016) | 8.686 (2.9493)
  2d-4h | 8.857 (2.5687) | 9.450 (3.1889)
  2d-8h | 10.471 (3.0698) | 9.064 (2.8527)
  2d-12h | 9.543 (3.5213) | 9.514 (3.6367)
  2d-16h | 9.343 (3.4469) | 8.821 (3.6413)
  2d-20h | 8.807 (3.4130) | 7.807 (2.8073)
  3d-0h | 8.135714 (2.5548166) | 8.250000 (4.3164711)
  3d-4h | 8.579 (2.8282) | 9.486 (3.7223)
  3d-8h | 9.121 (2.8011) | 8.879 (3.0238)
  3d-12h | 8.721 (2.8072) | 9.429 (3.0648)
  3d-16h | 9.328571 (3.2257208) | 8.935714 (2.2210902)
  3d-20h | 8.250000 (2.3299884) | 7.957143 (2.0129253)

6. Secondary Outcome: Length of Hospital Stay (LOS)
Description: every participators stayed in hospital
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Groups:
- Intermittent Feeding With Semi-solid Nutrients: intermittent feeding with semi-solid nutrients:after infusion of semi-solid agent, enteral nutrition is applied less than 60 mins.
  Intervention: Other: bolus Intermittent enteral feeding
  semi-solid agent: after infusion of semi-solid agent, Intermittent enteral feeding is applied less than 60 mins
Arm/Group | Intermittent Feeding With Semi-solid Nutrients | Intermittent Feeding
Number analyzed (Participants) | 14 | 14
days | 20.07 (25.71) | 14.36 (7.59)
Statistical Analysis 1: Comparison: Intermittent Feeding With Semi-solid Nutrients vs Intermittent Feeding; Test type: Non-Inferiority — According to the rule of a=0.05, P<0.05 means that the hypothesis was true; p < 0.05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Total follow-up 1 month
Groups:
- Standard Enteral Nutrition; Semi-solidification With Nutrient: We only record the daily enteral nutrition prescribed and received as well as the acute complications of enteral nutrition (EN) such as diarrhea, vomiting, regurgitation, bowel distension and lung infection in this study, no other adverse was found
Arm/Group | Standard Enteral Nutrition | Semi-solidification With Nutrient
All-Cause Mortality (participants affected / at risk) | 2/14 | 3/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT03017079/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT03017079/SAP_001.pdf
  • Informed Consent Form (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT03017079/ICF_002.pdf